CLINICAL TRIAL: NCT06061510
Title: Fish Oil-derived Omega-3 Fatty Acids on Gut Microbiota and Lipid Metabolome in Type 2 Diabetes Mellitus: a Randomized, Double-blind, Placebo-Controlled Clinical Trial
Brief Title: Fish Oil-derived Omega-3 Fatty Acids on Gut Microbiota and Lipid Metabolome in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Jia-yue Xia, Principal Investigator, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NO. 2019710-6
Record Dates: First submitted 2023-09-18; First posted 2023-09-29 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes Mellitus; Lipid Metabolism Disorder; Fatty Acid Metabolism Disorder
Keywords: Omega-3 Fatty Acids; Gut Microbiota; lipid Metabolome; glycerophospholipid; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Lipid Metabolism Disorders | interventions — Docosahexaenoic Acids; Corn Oil

STUDY DESIGN:
Intervention Model Description: The study was a randomised, double-blind trial.
Who Masked: Participant, Investigator
Masking Description: The study was a randomised, double-blind trial, and neither the subjects nor the research workers knew the exact subgroups or the progress of the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fish oil group (Experimental): Fish oil supplement capsules contained omega-3 polyunsaturated fatty acids supplied by Royal DSM Group, the Netherlands. Each 100 grams of fish oil capsules contains mainly 36.86 grams of EPA, 17.47 grams of DHA and other types of fatty acids.
  Interventions: Dietary Supplement: omega-3 polyunsaturated fatty acids
- The placebo group (Placebo Comparator): The placebo for fish oil contained corn oil (Each 100 grams of corn oil contained 45.64 grams of linoleic acid, 25.62 grams of oleic acid, 17.0 grams of palmitic acid, and other fatty acids).
  Interventions: Dietary Supplement: corn oil

INTERVENTIONS:
Dietary Supplement: omega-3 polyunsaturated fatty acids — Participants in the intervention group took fish oil capsules, 6 capsules per day, divided into two doses in the morning and two doses in the evening.
  Arms: fish oil group
Dietary Supplement: corn oil — Participants in the placebo group took corn oil capsules, 6 capsules per day, divided into two doses in the morning and two doses in the evening.
  Arms: The placebo group

SUMMARY:
The objective of this research was to investigate the impact of Omega-3 PUFAs on the gut microbiota and serum lipid metabolites in participants diagnosed with type 2 diabetes, employing high-throughput sequencing technology and untargeted lipidomics.

DETAILED DESCRIPTION:
The pathogenesis of diabetes is associated with perturbations in lipid metabolism and intestinal flora. Nevertheless, the precise impact of Omega-3 polyunsaturated fatty acids (Omega-3 PUFAs) on key lipid metabolites, intestinal microorganisms, and fungi linked to type 2 diabetes remains indeterminate. The objective of this research was to investigate the impact of Omega-3 PUFAs on the gut microbiota and serum lipid metabolites in participants diagnosed with type 2 diabetes, employing high-throughput sequencing technology and untargeted lipidomics. The investigators randomly allocated 110 eligible participants into either the fish oil intervention group or the placebo control group for a 3-month double-blind randomized intervention trial. Bacterial 16S rDNA, fungal diversity analysis of Internally Transcribed Spacer sequences (ITS) and untargeted lipidomics were used to investigate the effects of Omega-3 PUFAs on intestinal microbiota and serum lipid metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes have been diagnosed;
* Male or female aged 18-70 years;
* After listening to the project presentation, voluntarily participate in the study and sign an informed consent form.

Exclusion Criteria:

* Pregnant or lactating women;
* Poorly controlled diabetes, i.e. HbA1c>9%；
* Have taken omega-3 PUFAs-related supplements in the past six months；
* Taking lipid-lowering drugs or other drugs that affect blood lipid metabolism；
* Patients with severe diabetic complications, severe hypertension, combined with
* diseases of the heart, brain, liver, kidney, thyroid and hematopoietic system, psychosis；
* Patients with severe immune system disorders；
* Have special diets: vegetarians, weight managers, ketogenic test takers, etc；
* The attending physician deems the participant unsuitable

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-06-08 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Concentration of Serum triglycerides | 12 weeks
  physiological parameter
Concentration of total cholesterol | 12 weeks
  physiological parameter
Concentration of low-density lipoprotein cholesterol | 12 weeks
  physiological parameter
Concentration of high-density lipoprotein cholesterol | 12 weeks
  physiological parameter
weight in kilograms | 12 weeks
  physiological parameter
height in meters | 12 weeks
  physiological parameter
body mass index (BMI) | 12 weeks
  BMI=weight(kg)/height^2(m)
waist circumference | 12 weeks
  physiological parameter
hip measurement | 12 weeks
  physiological parameter
Systolic blood pressure | 12 weeks
  physiological parameter
Diastolic blood pressure | 12 weeks
  physiological parameter

SECONDARY OUTCOMES:
Number of Participants who take drugs | 12 weeks
  This indicator refers to the number of participants taking medication.
Incidence of diabetes complications | 12 weeks
  This indicator refers to the proportion of participants experiencing complications from diabetes.
Rate of smoking among participants | 12 weeks
  This indicator refers to the proportion of participants who smoke.

CONTACTS AND LOCATIONS:
Locations (1):
- Southeast university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No